CLINICAL TRIAL: NCT05494697
Title: A Phase 2 Randomized Open-Label Controlled Study to Evaluate the Efficacy and Safety of Ampligen in Combination With Standard of Care Versus SOC Alone Following First-Line Therapy in Subjects With Locally Advanced Pancreatic Adenocarcinoma
Brief Title: Ampligen Combined With SOC Versus SOC Alone Following First-Line Therapy in Subjects With LAPC
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: A business decision to place screening/enrollment on hold. Study redesign/amendment pending additional Ampligen-related data from an ongoing Phase I-II open label study (NCT05927142)
Sponsor: AIM ImmunoTech Inc. (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMP-270
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — poly(I).poly(c12,U)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ampligen / rintatolimod + SOC Chemoradiation (Experimental): Subjects will receive rintatolimod [intravenous (IV)], up to 400 mg twice weekly plus SOC chemoradiation until disease progression
  Interventions: Drug: Rintatolimod
- SOC Chemoradiation Alone (No Intervention): Subjects will receive SOC chemoradiation until evidence of disease progression.
- Ampligen / rintatolimod + SOC (Experimental): Subjects will receive rintatolimod [intravenous (IV)], up to 400 mg twice weekly plus SOC (SOC does not include chemoradiation) until disease progression
  Interventions: Drug: Rintatolimod
- SOC Alone (No Intervention): Subjects will receive SOC (SOC does not include chemoradiation) until evidence of disease progression.

INTERVENTIONS:
Drug: Rintatolimod — Rintatolimod (poly I : poly C12U)
  Other Names: Ampligen; poly I : poly C12U
  Arms: Ampligen / rintatolimod + SOC; Ampligen / rintatolimod + SOC Chemoradiation

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Ampligen in patients with locally advanced pancreatic adenocarcinoma

DETAILED DESCRIPTION:
This is a Phase 2, randomized, open-label controlled study to evaluate the efficacy and safety of Ampligen treatment combined with standard of care (SOC) versus SOC alone following First-line therapy in subjects with locally advanced pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of pancreatic adenocarcinoma confirmed pathologically: Unresectable pancreatic cancer; locally advanced pancreatic cancer.
2. Measurable disease per RECIST v.1.1.
3. Completion of at least four (4) months of first line therapy, such as FOLFIRINOX and no disease progression per RECIST v.1.1 as confirmed by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) scan after last first-line therapy and prior to randomization.
4. Subject must meet one of the following criteria for stratification question of 'Is subject planned to receive chemoradiation therapy as SOC? [Yes/No]' A. For subjects to be enrolled under stratification of 'Yes, SOC includes chemoradiation', subjects are planned to receive the following allowable radiotherapy and chemotherapy, with curative intent (i.e., not palliative).

   Allowable SOC radiotherapy:
   * IMRT (Intensity-Modulated Radiation Therapy)
   * SBRT (Stereotactic Body Radiation Therapy)

   Allowable SOC chemotherapy:
   * Capecitabine
   * 5-Fluorouracil (5-FU) +/- irinotecan B. For subjects to be enrolled under stratification of 'No, SOC does not include chemoradiation', subjects are planned to receive chemotherapy alone or undergo surveillance for disease progression only.
5. Male or non-pregnant, non-lactating female, ≥18 years or age.
6. Negative serum pregnancy test at screening visit for female subjects of childbearing potential. Females of childbearing potential must be willing to use an acceptable method of contraception from screening up until 90 days after last study treatment administration.

   Acceptable methods of contraception include abstinence, female subject/partner's use of hormonal contraceptive (oral, patch, injectable, depot or vaginal) in conjunction with a barrier method (e.g., diaphragm, cervical cap, condom, spermicide or sponge), or female subject/partner's use of an implantable device (implantable rod or intrauterine device).

   Female subject/partners of non-childbearing potential are defined as surgically sterile (e.g., bilateral tubal ligation, hysterectomy) or two years postmenopausal at time of screening.

   All male subjects (excluding men who have been sterilized) with female partners of child-bearing potential must agree to consistently and correctly use a condom from screening up until 90 days after last study treatment administration. In addition, subjects may not donate sperm for the same time period.
7. Provide signed written informed consent and willingness, ability to comply with study requirements.
8. Minimum weight of 40kg at screening.
9. Karnofsky Performance Status of 80 or higher at screening.
10. Subject must have a projected life expectancy of ≥ 3 months in the opinion of the Investigator.
11. Subject has adequate organ function by the following laboratory assessments at screening (after the last dose of first-line therapy treatment and prior to randomization):

Hematologic:

Platelets ≥ 100×10^9/L Hemoglobin ≥ 9.0 g/dL Absolute Neutrophil Count (ANC) ≥ 1.5×10^9/L WBC ≥ 3 x 10^9/L Neutrophil/Lymphocyte (N/L) ratio < 4.5

Hepatic:

AST/ALT ≤ 3×ULN (if liver metastases are present, ≤ 5×ULN) Alkaline phosphatase ≤ 2.0×ULN (if liver metastases are present, ≤ 5×ULN) Total bilirubin ≤ 1.5×ULN Albumin ≥ 3.0 g/dL

Renal:

Creatinine clearance ≥ 60 mL/min using the Cockcroft-Gault formula.

Coagulation:

PT, aPTT and INR within normal limits

Exclusion Criteria:

1. Diagnosis of islet neoplasm acinar cell carcinoma, non-adenocarcinoma (i.e., lymphoma, sarcoma), adenocarcinoma originating from the biliary tree, or cystadenocarcinoma.
2. Subjects who have surgically resectable locally advanced pancreatic adenocarcinoma following treatment with first-line therapy, such as FOLFIRINOX.
3. Subject has received prior treatment with Ampligen®.
4. Therapy with investigational drugs within 6 weeks of beginning study medication.
5. History of prior malignancy, except for adequately treated in situ cancer, basal cell, squamous cell skin cancer, or other cancers (e.g., breast, prostate) for which the subject has been disease-free for at least 3 years. Subjects with prior cancer that is adequately controlled per the judgement of the Investigator will not be excluded from the study.
6. Any serious medical condition, laboratory abnormality, psychiatric illness, or comorbidity that, in the judgment of the Investigator, would make the subject inappropriate for the study.
7. Serious systemic fungal, bacterial, viral, or other infection that is not controlled or requires intravenous (IV) treatment for infection(s).
8. Known history of positivity (regardless of immune status) for human immunodeficiency virus (HIV).
9. Known history of, chronic active, or active viral hepatitis A, B, or C infection
10. Clinically significant bleeding within 2 weeks prior to Randomization (e.g., gastrointestinal [GI] bleeding, intracranial hemorrhage).
11. Pregnant or lactating women.
12. Myocardial infarction within the last 6 months prior to Randomization, symptomatic congestive heart failure (New York Heart Association Classification > Class II), unstable angina, or unstable cardiac arrhythmia requiring medication.
13. Subjects with abnormal electrocardiogram (ECG) at screening with QTc interval >470 ms (calculated using both the Bazett's and Fridericia's corrections).
14. Clinically significant ascites defined as requiring ≥ 1 paracentesis every 2 weeks.
15. Major surgery, defined as any surgical procedure that involves general anesthesia and a significant incision (i.e., larger than what is required for placement of central venous access, percutaneous feeding tube, or biopsy), within 28 days prior to Randomization or anticipated surgery during the study period.
16. Prior history of receiving immune checkpoint inhibitors (anti-CTLA4, anti-PD1, anti-PD- L1).
17. Inability to return for scheduled treatment and assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Randomization until disease progression, death, or end of study up to 182 weeks
  PFS is defined as the time, in months, from date of randomization to date of the first documentation of definitive disease progression as per RECIST v1.1 and iRECIST (the initial progressive disease (PD)) or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | Randomization to death due to any cause, or end of study up to 182 weeks.
  OS is defined as patients who are alive at time of analysis
Overall Survival (OS) at 1 year | Randomization to death due to any cause.at 1 year
  OS is defined as the time from date of Randomization to death due to any cause.
Objective Response Rate (ORR) | Randomization until disease progression, death, or end of study up to 182 weeks
  ORR is defined as the proportion of subjects who achieve a Complete Response (CR) or Partial Response (PR) as assessed by RECIST v1.1 and iRECIST
Duration of Response (DoR) | Randomization until disease progression, death, or end of study up to 182 weeks
  DoR is defined as the time from the date of the first documentation of objective tumor response (CR or PR) to the date of the first documentation of objective tumor progression per RECIST v1.1 and iRECIST or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: David R Strayer, MD, Study Director — AIM ImmunoTech Inc.
Locations (3):
- United States (3):
  - Nebraska Medical Center, Omaha, Nebraska
  - Gabrail Cancer Center Research, Canton, Ohio
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El Haddaoui H, Brood R, Latifi D, Oostvogels AA, Klaver Y, Moskie M, Mustafa DA, Debets R, van Eijck CHJ. Rintatolimod (Ampligen(R)) Enhances Numbers of Peripheral B Cells and Is Associated with Longer Survival in Patients with Locally Advanced and Metastasized Pancreatic Cancer Pre-Treated with FOLFIRINOX: A Single-Center Named Patient Program. Cancers (Basel). 2022 Mar 8;14(6):1377. doi: 10.3390/cancers14061377. PMID 35326528